CLINICAL TRIAL: NCT05140135
Title: Effectiveness and Mechanisms of Recovery Oriented Cognitive Therapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The funds used to originally support the study were withdrawn.
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 844100
Record Dates: First submitted 2021-11-17; First posted 2021-12-01 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recovery Oriented Cognitive Therapy (CT-R) (Experimental): Therapists implement CT-R in weekly sessions for approximately 9 months while supported by a clinical supervisor. Therapists will have completed a supervised CT-R training case prior to the initiation of the randomized controlled trial. CT-R will focus on strengthening aspirations and focusing on activities that can bring about one's desired life. The therapist will use techniques to engage the patient in the adaptive mode, which involves activating cognitions, affects, motivation, and behaviors by engaging the individual in personally meaningful activities.
  Interventions: Behavioral: Recovery Oriented Cognitive Therapy (CT-R)
- Continued Usual Care (Active Comparator)
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: Recovery Oriented Cognitive Therapy (CT-R) — The CT-R that will be implemented in the present study will focus on strengthening aspirations and focusing on activities that can bring about one's desired life. In CT-R, clinicians use techniques to engage the patient in the adaptive mode, which includes cognitions, affects, motivation, and behaviors that are activated when the individual is engaged in personally meaningful activities.
  Arms: Recovery Oriented Cognitive Therapy (CT-R)
Other: Treatment as Usual — All patients enrolled in the study who are randomized to the continued care as usual condition will continue to receive the treatments from their physician/treatment team at the Community Mental Health Center; however, they will not receive the adjunctive CT-R treatment.
  Arms: Continued Usual Care

SUMMARY:
This study is evaluating the effectiveness of recovery oriented cognitive therapy (CT-R) for patients with schizophrenia/schizoaffective disorder. To evaluate CT-R, the investigators are conducting a randomized controlled trial with patients from community mental health centers. Participants will be randomized to the CT-R condition, in which the participants will receive approximately 9 months of CT-R as an adjunctive treatment to current medical treatment, or to the continued usual care control condition.

The primary outcome measure (positive, negative, and general psychopathology symptoms) as well as secondary measures (quality of life, self-esteem, social anhedonia, recovery, dysfunctional attitudes, resilience, internalized stigma, and hopelessness) will be measured at baseline, 4-5 months after the first therapy appointment, approximately 9 months after the first therapy appointment, and approximately 15 months after the baseline appointment.

DETAILED DESCRIPTION:
Background/Purpose: Despite effective medical treatment, many patients with psychotic illnesses experience poor long-term functional outcomes possibly due to certain psychosocial factors that can interfere with recovery. CT-R was developed to address these factors by leading the individual to substantive progress by addressing any obstacles and promoting a cognitive shift in their beliefs in their own personal and social efficacy. The goal of this study is to evaluate the effectiveness and mechanisms of CT-R as an adjunctive treatment for individuals with schizophrenia/schizoaffective disorder.

Population: Participants will include individuals currently receiving pharmacological treatment for schizophrenia or schizoaffective disorder. Therapist participants who have preliminary training in CT-R will be recruited as well to deliver the treatment. Therapists will first complete a training phase consisting of a workshop and approximately 3 months of group supervision while providing CT-R to 1 training case each.

Intervention: The CT-R that will be implemented in the present study will focus on strengthening aspirations and focusing on activities that can bring about one's desired life. In CT-R, clinicians use techniques to engage the patient in the adaptive mode, which includes cognitions, affects, motivation, and behaviors that are activated when the individual is engaged in personally meaningful activities.

ELIGIBILITY:
Inclusion Criteria:

* Patients: Between 18 and 65 years old with a diagnosis of schizophrenia or schizoaffective disorder, proficient in English, currently under the care of a physician and on medication for schizophrenia/schizoaffective disorder, and able to provide informed consent.
* Therapists: 25 years of age or above, licensed therapist, preliminarily trained in CT-R.

Exclusion Criteria:

* Patients: Medical comorbidities causing brain damage (e.g., stroke, dementia), significant suicidal risk/ideation requiring immediate referral or suicidal gesture.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) | Up to 15 months after the baseline appointment
  Assesses positive, negative, and general psychopathology symptoms associated with schizophrenia. Consists of 33 items each rated on a scale from 1 (absent) to 7 (extreme).

SECONDARY OUTCOMES:
Quality of Life Scale (QLS) | Up to 15 months after the baseline appointment
  Measures quality in life of individuals living with schizophrenia and functioning. Total scores range from 0-126. Lower scores indicate lower quality of life and functioning.
Revised Social Anhedonia Scale (RSAS) | Up to 15 months after the baseline appointment
  Questionnaire assessing attitudes and preferences related to spending time with other people. Total score ranges from 0 to 20. Higher scores indicate a preference to spend time alone.
Beck Hopelessness Scale (BHS) | Up to 15 months after the baseline appointment
  Questionnaire measuring the extent of positive and negative beliefs about the future. Total score ranges from 0 to 20. Higher scores indicate higher levels of hopelessness.
Dysfunctional Attitude Scale (DAS) | Up to 15 months after the baseline appointment
  Self-report measure assessing levels of dysfunctional attitudes. It consists of 7 subscales for a total of 40 items. Each item is rated on a scale from 1 (totally agree) to 7 (totally disagree).
Road to Recovery Scale - 10 (RRS-10) | Up to 15 months after the baseline appointment
  Measures multi-faceted areas of recovery. Each item is rated on a 1-5 scale. Total score is averaged across items and ranges from 1 to 5. Higher scores indicate more pro-recovery behaviors.
Beck Self-Esteem Scale - Short Form (BSES-SF) | Up to 15 months after the baseline appointment
  Assesses beliefs about the self and others' impressions of the self. The 10-item version of the scale consists of 10 bipolar adjectives rated on a 10-point scale (anchors are "very much" for 1 and 10; "average" for 5 and 6).
Internalized Stigma of Mental Illness Inventory-29 (ISMI-29) | Up to 15 months after the baseline appointment
  Self-report instrument designed to measure the overall strength of respondents' internalized stigma of mental illness among persons with psychiatric disorders. Total score ranges from 29-116. Higher scores indicate greater levels of internalized stigma.
Connor-Davidson Resilience Scale (CD-RISC) | Up to 15 months after the baseline appointment
  Self-report measure designed to assess resilience. It also differentiates between patients with schizophrenia and healthy controls. Total scores range from 0 to 100, with higher scores indicating greater resilience.

CONTACTS AND LOCATIONS:
Locations (1):
- Eirini Zoupou, Philadelphia, Pennsylvania, United States